CLINICAL TRIAL: NCT03925363
Title: A Mobile Application to Increase Physical Activity, a Randomized Controlled Study
Brief Title: A Mobile Application to Increase Physical Activity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Region Västerbotten (Other Government)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Anna Nordström, Associate Professor, Region Västerbotten
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VCC_LIFE-5
Record Dates: First submitted 2019-02-14; First posted 2019-04-24 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will be randomized 1:1 to the feedback-app or the blind-app
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): Participants will be given a mobile-app where they will get feedback from the device based on their physical activity (feedback app)
  Interventions: Device: Physical activity mobile-application
- Control (Sham Comparator): Participants will be given a mobile-app that does not give feedback back, but the app will register physical activity (blind app).
  Interventions: Device: Physical activity mobile-application

INTERVENTIONS:
Device: Physical activity mobile-application — The active group will be given the feedback app and the control group the blind app

SUMMARY:
A mobile application will be tested in elderly men and women that is randomized to an application (blind-app) that registers physical activity or an application (feedback-app) where participants in addition set goals for physical activity and gets feedback from the application when these goals are achieved. Participants are randomized in permuted blocks of 10 to the blind-app or feedback-app. The primary outcome is increased physical activity. Secondary outcomes include, cardiovascular disease, diabetes, death, dementia, cancer, falls and fractures.

DETAILED DESCRIPTION:
In this randomized controlled study, it will be tested if a mobile application can increase physical activity and reduce the risk of later non-communicable disease.

Participants include individuals that previously have been included in a health survey (Healthy aging initiative, NCT03312439), with a low registered physical activity. Low physical is defined according to WHOs definition, i.e. at least 150 minutes of physical activity per week. Individuals will diabetes will be investigated separately.

Individuals will be excluded that cannot walk for exercise, or if they have diseases that severely affects the ability to exercise. We will also seek participants from the general population to be included with only two inclusion criteria; having a smart phone and at least 18 years of age.

Participants the meet the inclusion criteria will be randomized to an application that only registers physical activity (blind-app) or an application where the participants will set appropriate goals for physical activity and get proper feedback from the app when these goals are reached (feedback-app). Both groups will have individualized information about proper physical activity. Randomization will be made using sealed envelopes in permuted blocks of 10. Randomization will be stratified on year of birth and sex.

The primary outcome will be increased physical activity after 6 months. Secondary outcomes include cardiovascular disease, death, dementia, falls and fractures, diabetes, and improved glucose control in those that already have diabetes. Secondary outcomes also include changes in cardiovascular risk factors, such as blood pressure, blood lipids and obesity. Interaction analysis will be performed to investigate if the effects are different in men and women, based on baseline physical activity and based on age.

Based on the results from the previous health survey the individuals have participated in, a power analyses has been conducted. The participants physical activity were registered using accelerometers. The mean steps taken per week was 48000 with a standard deviation of 22000 steps. With assumption that the feedback-app will increase physical activity by at least 15%, 164 individuals would be needed in each group with an alpha level of 0.05 and a power of 80%. For secondary outcome of cardiovascular disease or death, estimates were based on incidence of these outcomes in 3617 individuals that participated in the health survey. During a mean follow up time of 928 days, 221 participants was diagnosed with cardiovascular disease or died during follow up, and 128 were diagnosed with cardiovascular disease. If assuming that the mobil-application will result in 15% lower risk of these two outcomes in those randomized to the feedback-app, 597 and 1371 individuals would be needed in each group, respectively, with the same follow up time. The effects during follow up will be monitored each year of follow up through patient registers. Follow up time is scheduled to a maximum of 2 years. We estimate that we then would need 895 and 2156 individuals in each group due to the shorter follow up time compared to in the example above.

ELIGIBILITY:
Inclusion Criteria:

* Previous participants in healthy aging initiative.

Exclusion Criteria:

* Not able to walk or previous medical diagnoses that severely limits the possibility to exercise.

Ages: 70 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 4000 (Estimated)
Dates: Start 2019-08-25 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
Increased physical activity as measured by the mobile application in steps per day | 3 years (anticipated)
  Increased physical activity in steps per day during the intervention period.

SECONDARY OUTCOMES:
Incidence of myocardial infarction | 3 years
  Diagnoses of myocardial infarction will be tracked using national registers.
Incidence of diagnosed diabetes | 3 years
  Diabetes diagnoses or start of treatment for diabetes will be tracked using national registers.
Incidence of diagnosed fractures | 3 years
  Diagnosed fractures will be tracked using national registers.
Incidence of diagnosed dementia | 3 years
  Diagnosed dementia or start of treatment using dementia drugs will be tracked using national registers.
Number of participants with high blood pressure | 1 year (anticipated)
  Systolic and diastolic blood pressure will be assessed at baseline and later using a sphygmomanometer.
Number of participants with high blood lipids | 1 year (anticipated)
  Blood lipids (cholesterol, LDL-cholesterol, and triglycerides) will be analyzed at baseline and after 6 and 12 months at the department of chemistry.
Number of participants with high blood glucose | 1 year (anticipated)
  Blood glucose will be analysed at the departement of clinical chemistry at baseline and follow up.
Grade of obesity | 1 year (anticipated)
  Obesity will be assessed using a non-elastic measurement tape at the waist
Body weight | 1 year (anticipated)
  Body weight in kilogram measured by a digital scale.
Incidence of stroke | 3 years
  Diagnoses of stroke will be tracked using national registers.
Incidence of angina pectoris | 3 years
  Diagnoses of angina pectoris will be tracked using national registers.
Incident mortality | 3 years
  Death during follow up will be tracked using national registers.
Number of participants with high glycated hemoglobin | 1 year (anticipated)
  Glycated hemoglobin will be measured at baseline and follow up at the Department of clinical chemistry

IPD SHARING:
Plan to Share IPD: No